CLINICAL TRIAL: NCT07042685
Title: Phase II Trial of 5-Fluorouracil (5FU)-Based Therapy in Combination With Fruquintinib as First Line in Patients With Locally Advanced Unresectable or Metastatic Colorectal Cancer
Brief Title: Trial of 5-Fluorouracil (5FU)-Based Therapy in Combination With Fruquintinib in Patients With Locally Advanced Unresectable or Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00039815 (HMCC-GI25-001)
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colorectal Cancer (CRC)
Keywords: first line; CRC; metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Drug Therapy; HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 5FU-based chemotherapy (FOLFIRI or mFOLFOX6) with fruquintinib (Experimental): The trial includes a single treatment arm in which all enrolled patients receive a combination of 5-Fluorouracil (5FU)-based chemotherapy and fruquintinib. Patients are treated with either the FOLFIRI or mFOLFOX6 (FOLFIRI: folinic acid, 5FU, irinotecan; or mFOLFOX6: folinic acid, 5FU, oxaliplatin) regimen, both of which include 5-fluorouracil (5FU), leucovorin (LV), and either irinotecan or oxaliplatin, respectively. Fruquintinib is administered orally once daily for 21 days of each 28-day cycle. The initial three patients receive 4 mg of fruquintinib daily to assess safety; if no dose-limiting toxicities are observed, the dose is increased to 5 mg for subsequent patients. Treatment continues until disease progression, unacceptable toxicity, or patient withdrawal. After six months, patients with stable disease or better transition to a maintenance phase with 5FU and fruquintinib alone.
  Interventions: Drug: Fruquintinib Combined With Chemotherapy

INTERVENTIONS:
Drug: Fruquintinib Combined With Chemotherapy — The intervention in this trial involves administering a combination of 5FU-based chemotherapy and fruquintinib to patients with locally advanced unresectable or metastatic colorectal cancer. Patients receive either the FOLFIRI or mFOLFOX6 regimen, both of which include 5-fluorouracil (5FU), leucovorin (LV), and either irinotecan (FOLFIRI) or oxaliplatin (mFOLFOX6). Fruquintinib is given orally once daily for 21 days in each 28-day cycle. The initial dose of fruquintinib is 4 mg daily for the first three patients to assess safety; if no dose-limiting toxicities are observed, the dose is increased to 5 mg daily for subsequent participants. Treatment continues until disease progression, unacceptable toxicity, or patient withdrawal. After six months, patients with stable disease or better transition to a maintenance phase with 5FU and fruquintinib alone.
  Other Names: Fruquintinib

SUMMARY:
This Phase II clinical trial at Houston Methodist Neal Cancer Center is evaluating the safety and efficacy of combining 5-Fluorouracil (5FU) -based chemotherapy (either FOLFIRI: folinic acid, 5FU, irinotecan; or mFOLFOX6: folinic acid, 5FU, oxaliplatin) with fruquintinib as a first-line treatment for patients with locally advanced unresectable or metastatic colorectal cancer. Fifty patients will receive treatment in 28-day cycles, with fruquintinib initially dosed at 4 mg daily and potentially increased to 5 mg if no significant toxicities are observed. After six months, patients showing stable disease or better will transition to a maintenance phase with 5FU and fruquintinib, continuing until disease progression or other discontinuation criteria are met. The primary endpoint is time to progression based on RECIST v1.1 criteria, while secondary endpoints include safety, tolerability, and duration of response. The trial is being conducted across multiple Houston Methodist hospitals and is currently the only first-line CRC trial available in the system. If successful, it could offer a new therapeutic option and inform future treatment guidelines for advanced colorectal cancer.

DETAILED DESCRIPTION:
This is a phase II trial investigating the efficacy and safety of 5-Fluorouracil (5FU)-based therapy in combination with fruquintinib for patients with locally advanced unresectable or metastatic colorectal cancer in the first-line setting at Houston Methodist Neal Cancer Center. Patients will be administered 5FU-based therapy combined with fruquintinib. This study will consist of the 5FU-based therapy administered to 50 patients as FOLFIRI (Irinotecan: 180mg/ m² I.V. 30-90min day 1, LV: 400mg/ m² I.V. 2 hours day 1, 5FU: 400mg/ m² I.V. bolus day 1; 2400mg/ m² I.V. 46-48 hours, in 2 weeks cycle), or mFOLFOX6 (Oxaliplatin: 85mg/ m² I.V. 2 hours day 1, LV: 400mg/ m² I.V. 2hours day1, 5FU: 400mg/ m² I.V. bolus day 1; 2400mg/m 2 I.V. 46-48 hours, in 2 weeks cycle), and fruquintinib orally once daily on days 1-21.The first 3 patients will receive fruquintinib at 4 mg orally once daily of each cycle. If no dose-limiting toxicity (DLT)-like adverse events related to fruquintinib are observed during the first two cycles, then subsequent patients will be enrolled at 5 mg orally once daily. Both fruquintinib and 5FU-based therapy doses will be adjusted as needed according to the Principal Investigator's opinion. Treatments will be 28-day cycles until disease progression, unacceptable toxicity, or consent withdrawal. After six months on the trial treatment, patients who have stable disease, partial response or complete response will transition to maintenance therapy which consists of 5-FU and fruquintinib, continuing until disease progression, unacceptable toxicity, or consent withdrawal. Following the study treatment period, patients who maintain a favorable response will be offered to continue the trial regimen off-protocol. The total study duration is approximately 12 months which encompasses both the initial treatment phase (6 cycles/6months) and the maintenance phase. There is no pre-specified maximum duration for the maintenance phase; treatment will continue until disease progression, unacceptable toxicity, or patient withdrawal. This ensures that patients deriving clinical benefit from the therapy can continue treatment as long as it remains safe and effective.

The primary endpoint will be evaluating the time to progression (TTP) of the patient population according to RECIST v1.1 criteria. A secondary endpoint will be assessing the safety and tolerability of 5FU-based therapy in combination with fruquintinib, as measured through the incidence and severity of treatment-emergent AEs (NCI CTCAE (v5.0)) and change from baseline in the clinical laboratory and physical examination findings. All grades of adverse event rates will be assessed and reported. An additional secondary endpoint will be measuring the duration of response of 5FU-based treatment in combination with fruquintinib in a first-line setting for locally advanced unresectable or metastatic colorectal cancer patients according to RECIST v1.1 criteria and using the investigator's tumor assessment. This study will be conducted within the Houston Methodist System including the Neal Cancer Center with full access to the naïve treatment population at other Houston Methodist community hospitals such as Houston Methodist Baytown Hospital, Houston Methodist Sugar Land Hospital, Houston Methodist Willowbrook Hospital, Houston Methodist West Hospital, Houston Methodist Clear Lake Hospital, Houston Methodist Cypress Hospital, and other Houston Methodist locations. Outreach materials such as brochures, fact sheets, flyers, and posters with our trial information will be compiled and distributed to our Houston Methodist Neal Cancer Center and Health System colleagues. Automated follow-up emails or text messages will remind patients to take the next step with their providers.

This study has no competing trial active at the Houston Methodist System, including the Neal Cancer Center or other community hospitals, making this the only first-line CRC trial available. If successful, the proposed therapy will represent a new option, in the first-line setting, for the treatment of locally advanced unresectable or metastatic colorectal cancer. This single-arm study may provide insights that could inform future guidelines enabling studies to better treat and control CRC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Written informed consent is required before performing any trial-specific tests or procedures. Signing of the informed consent form can occur outside the 28-day screening period.
3. Histopathologically or cytologically confirmed locally advanced unresectable or metastatic colorectal cancer. The study will include an all-comer population, meaning that patients will not be excluded based on specific molecular markers such as microsatellite instability-high (MSI-H) or B-Raf proto-oncogene mutations (BRAF mutations). However, as part of the Standard of Care, comprehensive molecular testing will be performed to assess MSI status, and other relevant biomarkers. For patients with MSI-H or BRAF mutations confirmed, treatment may be adjusted per Standard of Care practices.
4. Measurable disease per RECISTv1.1.
5. No prior systemic treatment. Patients with resected disease who later develop unresectable recurrence without prior systemic therapy remain eligible.
6. ECOG performance status of 0 or 1.
7. Life expectancy ≥6 months per treating physician's assessment.
8. Patients of childbearing potential must agree to use an adequate method of contraception during the study and for 30 days after the last dose of study treatment.
9. Patients must be able to swallow oral tablets.

Exclusion Criteria:

1. Hematology laboratory values of:

   1. Absolute neutrophil count ≤1500 cells/mm3
   2. Platelets ≤100,000 cells/mm3
   3. Hemoglobin ≤9 g/dL
   4. White blood count ≤3000 cells/mm3.
2. Hepatic laboratory values of aspartate transaminase (AST) or alanine aminotransferase (ALT):

   1. >5 × upper limits of normal (ULN) if the documented history of hepatic metastases; or
   2. >2.5 × ULN if no liver metastases are present.
3. Serum albumin <2.8 g/dL.
4. Total bilirubin >1.7 mg/dL × ULN.
5. Prothrombin time (PT) or international normalized ratio (INR) >1.5 × ULN. Note: Patients receiving therapeutic doses of anticoagulant therapy may be considered eligible if PT and INR are within the acceptable institutional therapeutic limits.
6. Serum creatinine or serum urea >1.5 × ULN.
7. Estimated glomerular filtration rate <50 mL/min.
8. Urine dipstick or urinalysis with protein ≥2+ or 24-hour urine protein ≥1.0 g/24-h. Subjects with 1+ proteinuria must undergo a 24-hour urine collection to assess urine protein level.
9. Positive pregnancy test, pregnant, or breastfeeding for all women of child-bearing potential.
10. Per treating physician's assessment, any other clinically significant laboratory abnormality that would compromise patient safety or the outcome of the study.
11. Any clinically significant and/or uncontrolled cardiac-related abnormality that would compromise patient safety or the outcome of the study including, but not limited to:

    1. Arrhythmia
    2. Bradycardia
    3. Tachycardia
    4. Symptomatic valvular disease
    5. Symptomatic congestive heart failure is classified by the New York Heart Association as Class III or IV
    6. Unstable angina pectoris.
12. Myocardial infarction within the past 6 months from consent.
13. Active bleeding diathesis.
14. Current complaints of persistent constipation or history of chronic constipation, untreatable bowel obstruction, or fecaloma within the past 6 months from consent.
15. Receiving chronic treatment with corticosteroids ≥5 mg of prednisone per day (or equivalent) or other systemic immunosuppressive agents. Topical or nasal corticosteroids are allowed.
16. Known history and/or uncontrolled hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV)-1 or HIV-2.
17. History of galactose intolerance, deficiency of Lapp lactase, or glucose-galactose malabsorption.
18. History of malignancy or active treatment for malignancy other than CRC (i.e., radiation or chemotherapy, including monoclonal antibodies) within 5 years. Note: Patients with squamous or basal cell carcinomas of the skin, carcinomas in situ of the cervix or uterus, ductal breast cancer in situ, resected low-grade prostate cancer, or other malignancies that in the opinion of the investigator are considered cured may participate.
19. Receipt of live, attenuated vaccine (e.g., intranasal influenza, measles, mumps, rubella, varicella) or close contact with someone who has received a live, attenuated vaccine within the past 1 month from consent. Note: Influenza vaccine will be allowed if administered >21 days.
20. Receipt of any investigational agent or study treatment within the past 30 days from consent for a condition other than CRC.
21. Receipt of any protein or antibody-based therapeutic agents (e.g., growth hormones or monoclonal antibodies) within the past 3 months from consent for a condition other than CRC.
22. Uncontrolled hypertension
23. Active infection requiring treatment
24. Recent history of major surgery
25. Thromboembolic events during the past 6 months
26. Adults unable to consent
27. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Time to Progression of 5FU in combination with fruquintinib in first-line metastatic colorectal cancer patients | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws, whichever comes first, assessed up to 24 months.
  To assess the time to progression (TTP) of patients with locally advanced unresectable or metastatic colorectal cancer (mCRC) treated with 5-Fluorouracil (5FU)-based therapy in combination with fruquintinib, according to RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Incidence of toxicity of 5FU in combination with fruquintinib in first-line metastatic colorectal cancer patients | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws from the study, whichever came first, assessed up to 13 months.
  To assess the safety profile, toxicity (all grades of adverse event rates) of 5-Fluorouracil (5FU)-based therapy in combination with fruquintinib in patients with locally advanced unresectable or metastatic colorectal cancer (mCRC) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Duration of the response of 5FU in combination with fruquintinib in first-line metastatic colorectal cancer patients | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws, whichever comes first, assessed up to 24 months.
  To evaluate the duration of the response of 5-Fluorouracil (5FU)-based therapy in combination with fruquintinib in the first-line setting for locally advanced unresectable or metastatic colorectal cancer (mCRC) patients from onset of response to progression or death, whichever occurs earlier according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria and investigator's tumor assessment.

OTHER OUTCOMES:
Overall Survival rate of first-line metastatic colorectal cancer patients with 5FU in combination with fruquintinib | From date of initial treatment, 6 and 12 months, assessed up to 24 months until death.
  To evaluate the overall survival (OS) rate of patients with locally advanced unresectable or metastatic colorectal cancer (mCRC) treated with 5-Fluorouracil (5FU)-based therapy in combination with fruquintinib at 6 and 12 months.
Overall Response Rate of first-line metastatic colorectal cancer patients with 5FU in combination with fruquintinib | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws, whichever comes first, assessed up to 24 months.
  To evaluate the overall response rate (ORR), disease control rate (DCR) and progression-free survival (PFS) of patients with locally advanced unresectable or metastatic colorectal cancer (mCRC) treated with 5-Fluorouracil (5FU)-based therapy in combination with fruquintinib at 6 and 12 months.
Changes in health-related quality of life for first-line metastatic colorectal cancer patients with 5FU in combination with fruquintinib | From baseline to months 6 and 12
  Changes in health-related quality of life from baseline to months 6 and 12, as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The EORTC QLQ-C30 scores range from 0 to 100. For global health status/quality of life and functional scales (e.g., physical, role, emotional, cognitive, social), higher scores indicate better outcomes (improved quality of life or functioning). For symptom scales/items (e.g., fatigue, pain, nausea/vomiting), higher scores indicate worse outcomes (more severe symptoms).
Time to treatment failure of 5FU in combination with fruquintinib in first-line patients with metastatic colorectal cancer | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws from the study, whichever came first, assessed up to 24 months.
  The number of months from beginning of treatment to the time of progression of patients on 5-Fluorouracil (5FU)-based therapy in combination with fruquintinib for patients with locally advanced unresectable or metastatic colorectal cancer (mCRC).

CONTACTS AND LOCATIONS:
Overall Officials: Maen Abdelrahim, MD, PhD, Pharm D, Principal Investigator — The Methodist Hospital Research Institute; Abdullah Esmail, MD, Study Director — Houston Methodist Neal Cancer Center
Locations (1):
- Houston Methodist Neal Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The Clinical Study Report will include analysis of de-identified data and will be shared with the supporter and published when available.
Supporting Information: CSR

REFERENCES:
- [Background] Sawicki T, Ruszkowska M, Danielewicz A, Niedzwiedzka E, Arlukowicz T, Przybylowicz KE. A Review of Colorectal Cancer in Terms of Epidemiology, Risk Factors, Development, Symptoms and Diagnosis. Cancers (Basel). 2021 Apr 22;13(9):2025. doi: 10.3390/cancers13092025. PMID 33922197
- [Background] Biller LH, Schrag D. Diagnosis and Treatment of Metastatic Colorectal Cancer: A Review. JAMA. 2021 Feb 16;325(7):669-685. doi: 10.1001/jama.2021.0106. PMID 33591350
- [Background] Ferrara N. VEGF and the quest for tumour angiogenesis factors. Nat Rev Cancer. 2002 Oct;2(10):795-803. doi: 10.1038/nrc909. PMID 12360282
- [Background] Wilhelm SM, Dumas J, Adnane L, Lynch M, Carter CA, Schutz G, Thierauch KH, Zopf D. Regorafenib (BAY 73-4506): a new oral multikinase inhibitor of angiogenic, stromal and oncogenic receptor tyrosine kinases with potent preclinical antitumor activity. Int J Cancer. 2011 Jul 1;129(1):245-55. doi: 10.1002/ijc.25864. Epub 2011 Apr 22. PMID 21170960
- [Background] Bergers G, Song S, Meyer-Morse N, Bergsland E, Hanahan D. Benefits of targeting both pericytes and endothelial cells in the tumor vasculature with kinase inhibitors. J Clin Invest. 2003 May;111(9):1287-95. doi: 10.1172/JCI17929. PMID 12727920
- [Background] Apperley JF, Gardembas M, Melo JV, Russell-Jones R, Bain BJ, Baxter EJ, Chase A, Chessells JM, Colombat M, Dearden CE, Dimitrijevic S, Mahon FX, Marin D, Nikolova Z, Olavarria E, Silberman S, Schultheis B, Cross NC, Goldman JM. Response to imatinib mesylate in patients with chronic myeloproliferative diseases with rearrangements of the platelet-derived growth factor receptor beta. N Engl J Med. 2002 Aug 15;347(7):481-7. doi: 10.1056/NEJMoa020150. PMID 12181402
- [Background] Li J, Qin S, Xu RH, Shen L, Xu J, Bai Y, Yang L, Deng Y, Chen ZD, Zhong H, Pan H, Guo W, Shu Y, Yuan Y, Zhou J, Xu N, Liu T, Ma D, Wu C, Cheng Y, Chen D, Li W, Sun S, Yu Z, Cao P, Chen H, Wang J, Wang S, Wang H, Fan S, Hua Y, Su W. Effect of Fruquintinib vs Placebo on Overall Survival in Patients With Previously Treated Metastatic Colorectal Cancer: The FRESCO Randomized Clinical Trial. JAMA. 2018 Jun 26;319(24):2486-2496. doi: 10.1001/jama.2018.7855. PMID 29946728
- [Background] Dasari A, Lonardi S, Garcia-Carbonero R, Elez E, Yoshino T, Sobrero A, Yao J, Garcia-Alfonso P, Kocsis J, Cubillo Gracian A, Sartore-Bianchi A, Satoh T, Randrian V, Tomasek J, Chong G, Paulson AS, Masuishi T, Jones J, Csoszi T, Cremolini C, Ghiringhelli F, Shergill A, Hochster HS, Krauss J, Bassam A, Ducreux M, Elme A, Faugeras L, Kasper S, Van Cutsem E, Arnold D, Nanda S, Yang Z, Schelman WR, Kania M, Tabernero J, Eng C; FRESCO-2 Study Investigators. Fruquintinib versus placebo in patients with refractory metastatic colorectal cancer (FRESCO-2): an international, multicentre, randomised, double-blind, phase 3 study. Lancet. 2023 Jul 1;402(10395):41-53. doi: 10.1016/S0140-6736(23)00772-9. Epub 2023 Jun 15. PMID 37331369
- [Background] Mohelnikova-Duchonova B, Melichar B, Soucek P. FOLFOX/FOLFIRI pharmacogenetics: the call for a personalized approach in colorectal cancer therapy. World J Gastroenterol. 2014 Aug 14;20(30):10316-30. doi: 10.3748/wjg.v20.i30.10316. PMID 25132748
- [Background] Ishiguro M, Kotake K, Nishimura G, Tomita N, Ichikawa W, Takahashi K, Watanabe T, Furuhata T, Kondo K, Mori M, Kakeji Y, Kanazawa A, Kobayashi M, Okajima M, Hyodo I, Miyakoda K, Sugihara K. Study protocol of the B-CAST study: a multicenter, prospective cohort study investigating the tumor biomarkers in adjuvant chemotherapy for stage III colon cancer. BMC Cancer. 2013 Mar 25;13:149. doi: 10.1186/1471-2407-13-149. PMID 23530572
- [Background] Reddy TP, Khan U, Burns EA, Abdelrahim M. Chemotherapy rechallenge in metastatic colon cancer: A case report and literature review. World J Clin Oncol. 2020 Nov 24;11(11):959-967. doi: 10.5306/wjco.v11.i11.959. PMID 33312889
- [Background] Glimelius B, Stintzing S, Marshall J, Yoshino T, de Gramont A. Metastatic colorectal cancer: Advances in the folate-fluoropyrimidine chemotherapy backbone. Cancer Treat Rev. 2021 Jul;98:102218. doi: 10.1016/j.ctrv.2021.102218. Epub 2021 May 4. PMID 34015686
- [Background] Vogel A, Hofheinz RD, Kubicka S, Arnold D. Treatment decisions in metastatic colorectal cancer - Beyond first and second line combination therapies. Cancer Treat Rev. 2017 Sep;59:54-60. doi: 10.1016/j.ctrv.2017.04.007. Epub 2017 May 4. PMID 28738235
- [Background] Diez M, Teule A, Salazar R. Gastroenteropancreatic neuroendocrine tumors: diagnosis and treatment. Ann Gastroenterol. 2013;26(1):29-36. PMID 24714698
- [Background] Colucci G, Gebbia V, Paoletti G, Giuliani F, Caruso M, Gebbia N, Carteni G, Agostara B, Pezzella G, Manzione L, Borsellino N, Misino A, Romito S, Durini E, Cordio S, Di Seri M, Lopez M, Maiello E, Montemurro S, Cramarossa A, Lorusso V, Di Bisceglie M, Chiarenza M, Valerio MR, Guida T, Leonardi V, Pisconti S, Rosati G, Carrozza F, Nettis G, Valdesi M, Filippelli G, Fortunato S, Mancarella S, Brunetti C; Gruppo Oncologico Dell'Italia Meridionale. Phase III randomized trial of FOLFIRI versus FOLFOX4 in the treatment of advanced colorectal cancer: a multicenter study of the Gruppo Oncologico Dell'Italia Meridionale. J Clin Oncol. 2005 Aug 1;23(22):4866-75. doi: 10.1200/JCO.2005.07.113. Epub 2005 Jun 6. PMID 15939922
- [Background] Bartsch F, Eberhard J, Ruckert F, Schmelzle M, Lehwald-Tywuschik N, Fichtner-Feigl S, Gaedcke J, Oldhafer KJ, Oldhafer F, Diener M, Mehrabi A, Settmacher U, Becker T, Keck T, Friess H, Strucker B, Opitz S, Lemke J, Schnitzbauer A, Lang H; German ICC Collaboration Group. Repeated resection for recurrent intrahepatic cholangiocarcinoma: A retrospective German multicentre study. Liver Int. 2021 Jan;41(1):180-191. doi: 10.1111/liv.14682. PMID 32997886